CLINICAL TRIAL: NCT06166888
Title: A Phase Ia/Ib, Multicenter and Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of Anti-PD-1 and CD73 Bispecific Antibody AK131 in Patients With Advanced Solid Tumors
Brief Title: A Study of AK131 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK131-101
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK131 (Experimental): Subjects will receive AK131 via intravenously (IV) Q2W or Q3W, up to 2 years
  Interventions: Drug: AK131

INTERVENTIONS:
Drug: AK131 — AK131 is an anti-PD-1 and CD73 bispecific antibody

SUMMARY:
This is a phase Ia/Ib study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of AK131 in advanced solid tumor patients

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent.
2. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
3. Life expectancy ≥3 months.
4. Histologically or cytologically documented unresectable advanced or metastatic malignant tumor that has failed or intolerant of standard therapy, or for which no effective standard therapy is available.
5. Subject must have at least one measurable lesion according to RECIST Version1.1.
6. Adequate organ function.
7. Female subjects of childbearing potential and male subjects with female partners of childbearing potential must agree to use effective barrier methods of contraception during the study and for 120 days after last dose of study drug.

Exclusion Criteria:

1. Any malignancy other than the disease under study within the past 3 years except for radically cured local cancers.
2. Being involved in another clinical study, except for observational clinical studies or follow-up period of interventional studies.
3. Receipt of any anti-CD73 treatment.
4. Anticancer therapy within 4 weeks prior to the first dose of investigational product.
5. Experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
6. Subjects with spinal cord compression or active brain metastases, except for subjects with untreated and asymptomatic brain metastases or with stable brain metastases after treatment.
7. Subjects with pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
8. Subjects whose imaging shows that the tumor has invaded important blood vessels or the investigator judges that the tumor is very likely to invade important blood vessels and cause fatal bleeding during the study.
9. Toxicities of prior anticancer therapy have not resolved to ≤ Grade 1.
10. Patients with clinically significant cardio-cerebrovascular disease.
11. Active autoimmune diseases or history of autoimmune diseases that may relapse.
12. History of interstitial lung disease or noninfectious pneumonitis.
13. Major surgery, trauma,unhealed wound, ulcer or fracture within 4 weeks prior to first dose of investigational product.
14. Any condition that required systemic treatment with corticosteroids or other immunosuppressive agents within 14 days prior to the first dose of investigational product.
15. Receipt of live attenuated vaccines within 4 weeks prior to the first dose of investigational product.
16. Known allergy or reaction to any component of the AK131 formulation.
17. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation.
18. Any other conditions that, in the opinion of the Investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicities (DLTs) | During the first 4 weeks
  DLTs will be assessed during the first 4 weeks of treatment. DLTs are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the DLT observation period.
Number of subjects with adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of study drug
  AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
Serum PK concentration of AK131 | From first dose of study drug through 30 days after last dose of study drug
  Serum PK concentration of AK131 in individual subjects at different time points after AK131 administration
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of study drug through 30 days after last dose of study drug
  The immunogenicity of AK131 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs)
Objective response rate (ORR) | Up to approximately 2 years
  ORR is defined as the proportion of subjects with confirmed CR or confirmed PR (based on RECIST Version 1.1).
Disease control rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (based on RECIST Version 1.1).
Progression-free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression (based on RECIST Version 1.1) or death due to any cause, whichever occurs first.
Time to response (TTR) | Up to approximately 2 years
  TTR is defined as the time from the start of the treatment to the first objective tumor response observed for patients who achieved CR or PR (based on RECIST Version 1.1).
Duration of Response (DoR) | Up to approximately 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST Version 1.1) or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to approximately 2 years
  OS defined as the time from the first dose to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinming Yu, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No